CLINICAL TRIAL: NCT03993236
Title: Moderate-intensity Rosuvastatin Plus Ezetimibe Versus High-intensity Rosuvastatin for Target LDL-C Goal Achievement in Patients With Recent Ischemic Stroke: a Randomized Clinical Trial
Brief Title: Study on Rosuvastatin+Ezetimibe and Rosuvastatin for LDL-C Goal in Patients With Recent Ischemic Stroke
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Keun-Sik Hong (Other)
Collaborators: Ewha Womans University Seoul Hospital (Other); Severance Hospital (Other); Korea University Ansan Hospital (Other); Korea University Guro Hospital (Other); Myongji Hospital (Other); Seoul St. Mary's Hospital (Other); Samsung Medical Center (Other); Seoul National University Hospital (Other); Chung-Ang University Hosptial, Chung-Ang University College of Medicine (Other); Hallym University Medical Center (Other); Kyunghee University Medical Center (Other); Inje University Ilsan Paik Hospital (Other)
Responsible Party: Sponsor-Investigator, Keun-Sik Hong, Principal Investigator, Inje University
Organization: Inje University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ROSETTA-Stroke
Record Dates: First submitted 2019-06-17; First posted 2019-06-20 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Stroke, Ischemic
Keywords: Stroke, Ischemic; Rosuvastatin; Ezetimibe
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rosuvastatin/Ezetimibe 10/10mg (Experimental): The experimental group is orally administered with rosuvastatin 10 mg plus ezetimibe 10 mg combination once daily for 90 days.
  Interventions: Drug: Experimental: Rosuvastatin/Ezetimibe 10
- Rosuvastatin 20mg (Active Comparator): The comparator group is orally administered with rosuvastatin 20 mg single agent once daily for 90 days
  Interventions: Drug: Active Comparator: Rosuvastatin 20mg

INTERVENTIONS:
Drug: Experimental: Rosuvastatin/Ezetimibe 10 — * Rosuvastatin/Ezetimibe 10/10mg
  * orally administered once daily for 90 days
  Other Names: Rosuzet tab 10/10 mg
  Arms: Rosuvastatin/Ezetimibe 10/10mg
Drug: Active Comparator: Rosuvastatin 20mg — * Rosuvastatin 20mg
  * orally administered once daily for 90 days
  Other Names: Suvast tab 20mg
  Arms: Rosuvastatin 20mg

SUMMARY:
A randomized clinical trial for the comparison of the efficacy and safety of moderate-intensity rosuvastatin plus ezetimibe versus high-intensity rosuvastatin for target LDL-C goal achievement in patients with recent ischemic stroke

DETAILED DESCRIPTION:
The purpose of this study is to compare the efficiency and safety on the target LDL-C goal achievement between rosuvastatin 10 mg plus ezetimibe 10 mg (rosuvastatin/ezetimibe 10/10 mg) once daily versus rosuvastatin 20 mg once daily in patients with recent ischemic stroke.

The target LDL-C goal achievement rate in patients with recent ischemic stroke has not been well studied. In particular, no clinical studies have been conducted comparing the efficacy and safety of low-dose rosuvastatin plus ezetimibe with high-dose rosuvastatin single agent for achieving target LDL-C levels.

In this trial, the investigators aim to compare the efficacy of the target LDL-C achievement between rosuvastatin 10 mg plus ezetimibe 10 mg (rosuvastatin/ezetimibe 10/10 mg) and rosuvastatin 20 mg in patients with recent ischemic stroke.

For this trial, more than 292 patients (584 total) per group will be enrolled.

Subjects who were satisfied with the inclusion/exclusion criteria of this trial and who agreed to participate in the clinical trial in writing were randomly assigned to a 1:1 ratio in the experimental group (the low-dose combination of rosuvastatin plus ezetimibe) and comparator group (high-dose rosuvastatin).

The duration of administration of the drug for clinical trials is 90 days (±14 days), and the efficacy and safety evaluation parameters are compared with baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with recent ischemic stroke who meet both 1) and 2) criteria below. 1) Patients with acute ischemic stroke confirmed by DWI(diffusion-weighted imaging)

   This is satisfied by meeting at least one of the following two criteria:
   1. Patients who sustained stroke symptoms for more than 24 hours and had acute ischemic lesions on DWI.
   2. Patients with acute ischemic lesions in DWI who had improved symptoms within 24 hours.

      2) Patients with ischemic stroke within 90 days.
2. Statin therapy indicated according to the recommendations of the 2014 American Heart Association/American Stroke Association guidelines.

   This is accomplished by meeting at least one of the following three criteria:
   1. Patients with ischemic stroke due to arteriosclerosis and LDL-C ≥ 100 mg / dL. (Class I; Level of Evidence B)
   2. Patients with ischemic stroke due to arteriosclerosis and LDL-C <100 mg / dL. (Class I; Level of Evidence C)
   3. Patients who require statin therapy due to other associated atherosclerotic cardiovascular disease. (Class I; Level of Evidence A).
3. Patients without statin dose within 28 days before ischemic stroke.
4. Patients who measured baseline LDL-C levels after an ischemic stroke. This is satisfied by meeting at least one of the following two criteria:

   1. Patients who had a baseline LDL-C level before the onset of a recent ischemic stroke and started statin therapy.
   2. Patients hospitalized with acute ischemic stroke who had baseline LDL-C levels after initiation of statin therapy should meet both of the following conditions:

      1. Patients with LDL-C levels measured within 3 days after initiation of statin therapy
      2. Patients in whom randomization and administration of the study drug can be administered within 7 days after baseline LDL-C measurement.
5. Adults over 19 years.
6. Those who voluntarily agreed in writing to the trial.

Exclusion Criteria:

1. Planned vascular intervention before the end of trial
2. Significant hepatic dysfunction (Aspartate Aminotransferase or Alanine Aminotransferase >120 IU/L)
3. Allergy or contraindication to rosuvastatin or ezetimibe
4. Alcohol or drug addiction
5. Pregnancy or breast-feeding
6. Severe anemia: Hb level <10 g/dL for men and <9 g/dL for women
7. Bleeding diathesis: platelet count <100,000/μl or prothrombin time International Normalized Ratio > 1·7
8. Inability or unwillingness to comply with study-related procedures
9. Employees of the investigator or study center, with direct involvement in the current study
10. Women unwilling to continue contraception during the study period
11. Participation in other clinical trials within three-month
12. Malignancy or other serious medical conditions with a life expectancy <6 months
13. Treatment with protease inhibitors or cyclosporine
14. Patients with severe renal impairment (creatinine clearance <30 mL / min)
15. Other reasons for ineligibility judged by investigators

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 584 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2021-09-27 (Actual); Study Completion 2021-09-27 (Actual)

PRIMARY OUTCOMES:
The percentage of subjects with LDL-C decreased more than 50% at 90days (±14 days) compared to Baseline | Baseline, Visit 4(Day 90)
  The percentage of subjects with LDL-C decreased more than 50% at 90days (±14 days) compared to Baseline

SECONDARY OUTCOMES:
Percentage of subjects with LDL-C less than 70 mg/dL at 90 days(±14 days) | Baseline, Visit 4(Day 90)
  Percentage of subjects with LDL-C less than 70 mg/dL at 90 days(±14 days)
The percentage of subjects with LDL-C decreased more than or less than 70 mg/dL at 90 days(±14 days) | Baseline, Visit 4(Day 90)
  The percentage of subjects with LDL-C decreased more than or less than 70 mg/dL at 90 days(±14 days)
The decrement of LDL-C at 90 days (±14 days) compared to baseline LDL-C (absolute difference and change) | Baseline, Visit 4(Day 90)
  The decrement of LDL-C at 90 days (±14 days) compared to baseline LDL-C (absolute difference and change)
The percentage of subjects achieved multiple lipid level (Total-C < 200mg/dL, LDL-C < 70mg/dL and triglyceride < 150mg /dL) | Baseline, Visit 4(Day 90)
  The percentage of subjects achieved multiple lipid level (Total-C < 200mg/dL, LDL-C < 70mg/dL and triglyceride < 150mg /dL)
Cardiovascular event rates including stroke (ischemic or hemorrhagic), coronary artery(myocardial infarction or coronary vascular reperfusion) and death related to vascular disease. | Baseline to Visit 4(up to 90 days)
  Cardiovascular event rates including stroke (ischemic of hemorrhagic), coronary artery(myocardial infarction or coronary vascular reperfusion) and death related to vascular disease.
Number of Death of all causes. | Baseline to Visit 4(up to 90 days)
  Number of Death of all causes.
Number of subjects with newly diagnosed diabetes. | Visit 4(Day 90)
  Number of subjects with newly diagnosed diabetes.
Fatigue scale measured by Fatigue Severity Scale. | Screening, Visit 4(Day 90)
  Fatigue scale measured by Fatigue Severity Scale. (The Fatigue Severity Scale is a 9-item scale which measures the severity of fatigue and its effect on a person's activity and lifestyle in patients with a variety of disorders. A 9-item questionnaire with questions related to how fatigue interferes with certain activities and rates its severity. The Fatigue Severity Scale scores range from 9 to 63, with higher scores indicating a greater fatigue severity.)
Incidence of rhabdomyolysis | Baseline to Visit 4(up to 90 days)
  Incidence of rhabdomyolysis
Incidence of serious liver dysfunction | Baseline to Visit 4(up to 90 days)
  Incidence of serious liver dysfunction (AST or ALT increase more than three times from baseline)

CONTACTS AND LOCATIONS:
Overall Officials: Keun-Sik Hong, MD., PhD., Principal Investigator — Department of Neurology, Inje University Ilsan Paik Hospital
Locations (12):
- South Korea (12):
  - Korea University Ansan Hospital, Ansan-si, Gyeonggi-do
  - Hallym University Medical Center, Anyang-si, Gyeonggi-do
  - Myongji Hospital, Goyang-si, Gyeonggi-do
  - Inje University Ilsan Paik Hospital, Ilsan, Gyeonggi-do
  - Chung-Ang University Hopital, Seoul
  - Ewha Womans University Seoul hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Kyung-Hee University Medical Center, Seoul
  - Samsung Medical Center, Sungkyunkwan University School of Medicine, Seoul
  - Seoul National University Hospital, Seoul
  - Seoul St Mary's Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hong KS, Bang OY, Park JH, Jung JM, Lee SH, Song TJ, Nam HS, Park HK, Jung KH, Heo SH, Koo J, Yu KH, Park KY, Kim CK, Park HK, Lee J, Lee J, Seo WK. Moderate-Intensity Rosuvastatin Plus Ezetimibe Versus High-Intensity Rosuvastatin for Target Low-Density Lipoprotein Cholesterol Goal Achievement in Patients With Recent Ischemic Stroke: A Randomized Controlled Trial. J Stroke. 2023 May;25(2):242-250. doi: 10.5853/jos.2022.02957. Epub 2023 Apr 11. PMID 37032475
- See also: publication — https://pubmed.ncbi.nlm.nih.gov/37032475/